CLINICAL TRIAL: NCT04638569
Title: Comparison of Obturator Nerve Block With Ultrasound Guidance and Anatomical Signs in Patients Undergoing Transurethral Resection
Brief Title: Comparison of Obturator Nerve Block With Ultrasound Guidance and Anatomical Signs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Eylem Yaşar, medical doctor of anesthesiology special, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 27/12/2019-19/VIII
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Succesful Obturator Nerve Block; Bladder Tumor; Bleeding
Keywords: obturator nerve block; bladder tumor; ultrasonografi; anatomical signs
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hemorrhage

STUDY DESIGN:
Intervention Model Description: group 1; Ultrasound-guided obturator nerve block group 2; obturator nerve block with anatomical signs
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided obturator nerve block group (Active Comparator): The ultrasound probe will be placed in the middle of the tuberculum pubis and femoral artery, 5-6 cm below the inguinal ligament, and 5 mL of 0.5% bupivacaine will be injected into the anterior and posterior branches of the ON with a needle.
  Interventions: Procedure: obturator nerve block
- obtutaror nerve block with anatomical landmarks (Active Comparator): In the second group, after the patient is placed in the lithotomy position, 1.5 cm lateral tuberculum pubis and 1.5 cm caudal will be marked and needle entry will be made and 0.5% bupivacaine will be injected with 10 mL.
  Interventions: Procedure: obturator nerve block

INTERVENTIONS:
Procedure: obturator nerve block — The ultrasound probe will be placed in the middle of the tuberculum pubis and femoral artery, 5-6 cm below the inguinal ligament, and 5 mL of 0.5% bupivacaine will be injected into the anterior and posterior branches of the ON with a needle. In the second group, after the patient is placed in the lithotomy position, 1.5 cm lateral tuberculum pubis and 1.5 cm caudal will be marked and needle entry will be made and 0.5% bupivacaine will be injected with 10 mL. The time elapsed until the first needle insertion and local anesthetic injection is completed will be recorded as the application time.

SUMMARY:
Comparison of the obturator nerve block in patients undergoing transurethral resection due to bladder tumor, technically using ultrasound guided or blinded with anatomical signs.

DETAILED DESCRIPTION:
The primary aim of this study is to compare the success rates of ONB techniques performed with ultrasound guided or blind technique. Its secondary purpose is to compare the effect of peroperative bleeding and control cystoscopy performed in the postoperative 3rd month on the presence of recurrent tumor.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients

Exclusion Criteria:

* Tumors that disrupt the integrity of the bladder,
* bladder floor tumors,
* coagulation disorders,
* motor in the lower limbs
* with sensory disturbances,
* uncooperative patients,
* Known allergy to local anesthetics
* patients with localized infection at the procedure site

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative succesful obturator nerve block | operation time
  peroperative adductor muscle spazm

SECONDARY OUTCOMES:
peroperative bleeding, Presence of recurrent tumor at postoperative 3rd month | 3 months
  peroperative bledding, Control by cystoscopy in the postoperative 3rd month recurrence tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Yaşar, Principal Investigator — Muğla Sıtkı Koçman University; Ali İhsan Uysal, Study Chair — Mugla Sitki Kocman University Department of Anesthesia; İlker Akarken, Study Chair — Mugla Sitki Kocman University Department of Urology; basak altiparmak, Study Chair — Mugla Sitki Kocman University Department of Anesthesia; semra demirbilek, Study Chair — Mugla Sitki Kocman University Department of Anesthesia
Locations (1):
- Mugla Sitki Kocman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No